CLINICAL TRIAL: NCT05706545
Title: Micro- and Macro-Circulation in Cardiac Surgery Patients
Acronym: MiMaC
Status: Suspended | Type: Observational
Why Stopped: Due to some problems in instrumentation acquisition the project has been currently suspended.
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Vlasta Bari, Assistant Professor, PhD, IRCCS Policlinico S. Donato
Other Study IDs: MiMaC
Record Dates: First submitted 2023-01-23; First posted 2023-01-31 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Surgery; Coronary Artery Bypass Graft; Surgical Aortic Valve Replacement
Keywords: autonomic nervous system; heart rate variability; cardiac surgery; major morbidities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Acquisition of cardiovascular signals and microcirculation sidestream darkfield images — ECG, arterial pressure and peripheral flow velocity via a percutaneous laser doppler will be acquired together with images of the sublingual microcirculation detected with sidestream darkfield images microscope

SUMMARY:
The hypothesis under the study is that there could be a link between a dysfunction in peripheral microcirculation, sublingual microcirculation or cardiovascular control and the development of post cardiac surgery major morbidities (stroke, acute kidney injury, prolonged intubation, mediastinitis, surgical reopening, death).

The state of sublingual microcirculation, of peripheral microcirculation and cardiovascular control will be assessed in 100 patients undergoing cardiac surgery during general anesthesia before the intervention and at the end of the intervention at the arrival in post-surgery ICU by means of signal processing techniques.

The extracted markers will be used to assess a statistical prediction model of major morbidities.

ELIGIBILITY:
Inclusion Criteria:

* age >18 yrs
* indication for a cardiac surgery intervention
* spontaneous sinus rhythm
* informed consent

Exclusion Criteria:

* know autonomic nervous systems pathologies or dysfunctions
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 consecutive patients scheduled for major cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2027-01 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Prediction of major morbidities by means of the variability of cardiovascular and hemodynamics markers | 24 months
  Statistical model assessment; time series variability analysis

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: No